CLINICAL TRIAL: NCT04913428
Title: Comparison of Blow-bottle Technique and Interdigital Breathing for Pulmonary Function of Post-laparotomy Patients .
Brief Title: Breathing Exercises for Pulmonary Function of Post-laparotomy Patients .
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00313 Huda Anjum
Record Dates: First submitted 2021-05-30; First posted 2021-06-04 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-05

CONDITIONS: Laparotomy Patients
Keywords: Pulmonary function; Chest expansion; Laparotomy; Spirometry

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interdigital exercise group (Experimental): Interdigital exercises:
  12 repetitions in 3 sets of 4 repetitions
  Conventional Physical Therapy:
  Incentive spirometer 3 - 4 times a day, Percussion twice a day, Mobilization of the patient Total session given was for 20 -30 minutes
  Interventions: Other: Interdigital exercise
- Blow-Bottle technique group (Active Comparator): Blow-Bottle technique:
  12 repetitions in 3 sets of 4 repetitions
  Conventional Physical Therapy:
  Incentive spirometer 3 - 4 times a day, Percussion twice a day, Mobilization of the patient Total session given was for 20 -30 minutes
  Interventions: Other: Blow-Bottle technique

INTERVENTIONS:
Other: Interdigital exercise — Patient asked to sit in upright position interlocking their fingers with inhaling deeply bringing the arms up and exhaling through mouth while bring the arm down.
  Arms: Interdigital exercise group
Other: Blow-Bottle technique — For blow bottle 20cm of bottle filled with 10cm of water in which a tube of length 35- 40cm inserted with the inner diameter of ≥8mm(21).Patient is asked to form bubbles in bottle by exhaling in bottle performing Forced Expiratory Techniques.
  Arms: Blow-Bottle technique group

SUMMARY:
The study is designed to compare the effects of blow bottle technique and interdigital exercises on the pulmonary functions of the post laparotomy patients where there is sudden decline in lung function and increased rate of complications after the surgery. A randomized control trial was conducted including post laparotomy patients, randomly allocated to interventional and control groups. Both the groups received breathing exercises along with conventional treatment during phase I rehabilitation. Data was collected at baseline, before and after every session and after 6 sessions before patient discharge from hospital. Outcome measures include assessment of lung volumes and capacities, oxygen saturation and vitals of the post laparotomy patients

DETAILED DESCRIPTION:
Pulmonary complications are common in post laparotomy patients because of multiple pre operative, intra operative and post operative factors. To manage these complications many interventions and breathing techniques are used. These complications alter the pulmonary function leading to decreased chest expansion, oxygen saturation and post operative atelectasis. Anesthetic drugs that also cause cardiac depression along with hemodynamic instability of the patient. Incision given to the chest or abdominal wall during procedure causes to lose the integrity of respiratory muscles which effects the functions of the muscle directly. Respiratory muscles are compromised, normal lung volumes are depressed. More than 75% of patients who are receiving neuromuscular blocking agent develops atelectasis. The estimated time after surgery for patient to return to its preoperative health status is approximately 6 weeks. These complications increase the hospital length of stay and cost associated with it as well as increase the morbidity and mortality.

Lung expansion techniques (LETs) are widely used to prevent postoperative pulmonary complications (PPCs). However, the effects of each of these techniques on thoraco-abdominal mechanics and PPC incidence after abdominal surgery remain unclear. Active Cycle of Breathing Techniques (ACBT) has shown to be effective in mobilizing and clearing the excess bronchial secretions and to improve lung function. It neither causes nor increases hypoxemia or increases airflow obstruction. Chest physiotherapy and breathing exercises are often prescribed to patients undergoing cardiac surgery and abdominal surgery in order to prevent or reduce post-operative pulmonary complications. There are different breathing techniques with and without mechanical devices after the surgery, but there is controversy regarding which breathing techniques are the most effective.

Researches have proved change in pulmonary functions by the use of various breathing exercises. Depressed pulmonary functions i.e. decreased forced vital capacity (FVC) , decreased forced expiratory volume (FEV1), Peak Expiratory Flow Rate (PEFR) are seen as result of disturbed lung function. Alteration in function of diaphragm contributes in postoperatively pulmonary function disturbances. Chest physiotherapy is implied for minimizing the altered lung functions and complications. This includes multiple breathing exercises, percussion , vibrations, huffing, coughing techniques, postural drainage and mobilization.

The current study is conducted to compare two respiratory techniques for the improvement in post operative pulmonary function; because of incisional pain, patients find the inspiratory exercises difficult to perform, therefore, the study is conducted to assess if easy-to -perform expiratory techniques are similar in effect to the inspiratory techniques and for the said purpose comparison of blow bottle technique and interdigital breathing on post laparotomy patients is made for the improvement of pulmonary function and vitals of these patients.

.

ELIGIBILITY:
Inclusion Criteria:

* Post laparotomy patients
* Age 25 to 45 years.
* Both genders.

Exclusion Criteria:

* Vitally unstable patients
* Complicated laparotomies
* Patients with post-operative complications e.g. delirium

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2018-09-20 (Actual)

PRIMARY OUTCOMES:
Peak expiratory flow rate (PEFR) | 5 days
  Peak expiratory flow rate (PEFR) measured through digital spirometer. Peak Expiratory Flow Rate (PEFR) measured through digital spirometer. Three zones of measurement are commonly used to interpret peak flow rates. Normal value of PEFR is (80-100%). Green zone indicates 80 to 100 percent of the usual or normal peak flow reading, yellow zone indicates 50 to 79 percent of the usual or normal peak flow readings, and red zone indicates less than 50 percent of the usual or normal peak flow readings.
Forced vital capacity (FVC) | 5 days
  Forced vital capacity (FVC) measured through digital spirometer. If the value of FVC is within 80% of the reference value, the results are considered normal.
Forced expiratory volume in 1sec (FEV1) | 5 days
  Forced expiratory volume in 1sec (FEV1) measured through digital spirometer. If the value of FEV1 is within 80% of the reference value, the results are considered normal.
FVC/FEV1 | 5 days
  FVC/FEV1 measured through digital spirometer. The normal value for the FEV1/FVC ratio is 70% (and 65% in persons older than age 65).

SECONDARY OUTCOMES:
Oxygen Saturation (SPO2) | 5 days
  Oxygen saturation measured through pulse oximeter as part of vitals
Heart rate | 5 days
  Heart rate is measured as part of vitals through heart rate monitor.
Chest expansion | 5 days
  Chest expansion at xiphoid level measured by finding the difference in measurements during inhalation and exhalation.
Respiratory rate | 5 days
  Respiratory rate calculated standing at bedside of patient.

CONTACTS AND LOCATIONS:
Overall Officials: Suman Sheraz, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Rawalpindi, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giacalone PL, Daures JP, Vignal J, Herisson C, Hedon B, Laffargue F. Pfannenstiel versus Maylard incision for cesarean delivery: A randomized controlled trial. Obstet Gynecol. 2002 May;99(5 Pt 1):745-50. doi: 10.1016/s0029-7844(02)01957-9. PMID 11978282
- [Background] Miskovic A, Lumb AB. Postoperative pulmonary complications. Br J Anaesth. 2017 Mar 1;118(3):317-334. doi: 10.1093/bja/aex002. PMID 28186222
- [Background] Dagan Y, Wiser I, Weissman O, Farber N, Hundeshagen G, Winkler E, Kazula-Halabi T, Haik J. An Improvised "Blow Glove" Device Produces Similar PEP Values to a Commercial PEP Device: An Experimental Study. Physiother Can. 2014 Summer;66(3):308-12. doi: 10.3138/ptc.2013-31. PMID 25125786
- [Background] Alaparthi GK, Augustine AJ, Anand R, Mahale A. Comparison of Diaphragmatic Breathing Exercise, Volume and Flow Incentive Spirometry, on Diaphragm Excursion and Pulmonary Function in Patients Undergoing Laparoscopic Surgery: A Randomized Controlled Trial. Minim Invasive Surg. 2016;2016:1967532. doi: 10.1155/2016/1967532. Epub 2016 Jul 21. PMID 27525116
- [Background] Craig DB. Postoperative recovery of pulmonary function. Anesth Analg. 1981 Jan;60(1):46-52. No abstract available. PMID 7006464
- [Background] Agostini P, Naidu B, Cieslik H, Steyn R, Rajesh PB, Bishay E, Kalkat MS, Singh S. Effectiveness of incentive spirometry in patients following thoracotomy and lung resection including those at high risk for developing pulmonary complications. Thorax. 2013 Jun;68(6):580-5. doi: 10.1136/thoraxjnl-2012-202785. Epub 2013 Feb 21. PMID 23429831
- [Background] Tyson AF, Kendig CE, Mabedi C, Cairns BA, Charles AG. The effect of incentive spirometry on postoperative pulmonary function following laparotomy: a randomized clinical trial. JAMA Surg. 2015 Mar 1;150(3):229-36. doi: 10.1001/jamasurg.2014.1846. PMID 25607594
- [Background] Lunardi AC, Paisani DM, Silva CCBMD, Cano DP, Tanaka C, Carvalho CRF. Comparison of lung expansion techniques on thoracoabdominal mechanics and incidence of pulmonary complications after upper abdominal surgery: a randomized and controlled trial. Chest. 2015 Oct;148(4):1003-1010. doi: 10.1378/chest.14-2696. PMID 25973670
- [Background] Westerdahl E, Lindmark B, Almgren SO, Tenling A. Chest physiotherapy after coronary artery bypass graft surgery--a comparison of three different deep breathing techniques. J Rehabil Med. 2001 Mar;33(2):79-84. doi: 10.1080/165019701750098920. PMID 11474953